CLINICAL TRIAL: NCT00229320
Title: Short Term Group Therapy for OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SHEBA-05-3679-JZ-CTIL
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Group therapy

SUMMARY:
Assessing OCD before and after group therapy

ELIGIBILITY:
Inclusion Criteria:

* OCD
* Eligibility to participate in group therapy

Exclusion Criteria:

* PTSD
* Suicidal thoughts
* Psychotic state
* Severe hostile personality disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Tel Aviv University
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel